CLINICAL TRIAL: NCT05489900
Title: Immunomodulatory Effect of Dexmedetomidine as an Adjuvant Drug in Laparoscopic Cholecystectomies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Gustavo N Silva, MD, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 50311621.0.0000.5258
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Physiological Effects of Drugs
Keywords: Immunomodulation; Dexmedetomidine; videolaparoscopic cholecystectomy
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients with Physical Health Status Classification 1 and 2, submitted to elective videolaparoscopic cholecystectomy surgery and previously signed the Free and Informed Consent Form. Continuous infusions of dexmedetomidine or 0.9% saline (placebo) were used in 52 patients. Dexmedetomidine was infused in the intervention group (26 patients) as follows: beginning of anesthetic induction after obtaining venous access at 1mcg/kg/h for 20 minutes, followed by 0.2 - 0.5 mcg/kg/h until the closure of the surgery. The placebo group (26 patients) received 0.9% saline infusion at the same rates as the intervention group.
Who Masked: Participant
Masking Description: Patients were randomly divided into two groups using the sequential distribution procedure of Pocock and Simon to balance the amount of sex and age group of patients between the groups. Participants' registration data were replaced by codes for the preservation of personal information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.9% Saline Infusion (No Intervention): The placebo group will receive 0.9% saline infusion at the same rates as the intervention group.
- Dexmedetomidine Infusion (Experimental): Dexmedetomidine will be used in the intervention group as follows: beginning in anesthetic induction after obtaining venous access at 1mcg/kg/h for 20 minutes, followed by 0.2 - 0.5 mcg/kg/h until the end of the surgery.
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine is a specific and potent α2-adrenergic agonist. By acting directly on the sympathetic nervous system, they can exert beneficial effects on the immune system through neuroimmune interactions. Its administration can induce an anti-inflammatory response due to different central (increase parasympathetic tone, promoting control of the inflammatory condition) and peripheral effects (stimulating innate immunity).(MILLER, 2015).
  Venous blood samples were collected at three times (T1, T2 and T3): Before anesthetic induction with collection in the preoperative environment on the day of surgery or during venoclysis before anesthetic induction (sample 1, T1); 6 hours after starting orifice closure and completion of drug or placebo infusion (sample 2, T2); and the last blood sample will be collected by me on the morning after the postoperative period, close to hospital discharge - 24h (sample 3, T3).
  Arms: Dexmedetomidine Infusion

SUMMARY:
Trauma triggers a tissue response involving the central nervous system, the hypothalamic-pituitary-adrenal axis and the immune system. There are many surgical and anesthetic factors that affect the response to trauma, and the control of the inflammatory factor is considered the most important. (KÜÇÜKEBE, O.B. ET AL, 2017). Dexmedetomidine is a specific α2-adrenergic agonist. By direct action on the sympathetic nervous system, α2-adrenergic agonists can exert beneficial effects on the immune system through neuroimmune interactions. Its administration can induce an anti-inflammatory response due to different central (increase parasympathetic tone, promoting control of the inflammatory condition) and peripheral effects (stimulating innate immunity). (MILLER, 2015). This study aims to evaluate the effect of dexmedetomidine administration in association with general anesthesia in a medium-sized surgical model, videolaparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The present study is a randomized, single-blind, prospective clinical trial. Its objective is to evaluate the possible qualitative changes in organic function and in the systemic inflammatory response when using dexmedetomidine associated with general anesthesia for laparoscopic cholecystectomy surgeries. The study was designed and executed according to the surgical routine of the Hospital Universitário Gaffré e Guinle - RJ. The anesthesiology service is recognized by the Ministry of Education and the Brazilian Society of Anesthesiology. Participant registration data will be replaced by codes for the preservation of personal information. The following were used in the elaboration of the study: 1) Selection of ASA I and II patients listed for elective procedures and standardization of the anesthetic technique. 2) A standardized data collection system in a specific form and fed with the residents with adequate supervision; 3) procedures converted into open surgery were excluded, since they imply an increase in surgical trauma and absence of pneumoperitoneum perfusion-reperfusion syndrome;4) Two groups with similar characteristics were used and the only difference will be the administration or not of dexmedetomidine in the procedure under study;5) Study with single blinding: the patient, also called the object of study, does not know which group he belongs to. The investigator does. Continuous infusions of dexmedetomidine or 0.9% saline (placebo) were used. Dexmedetomidine was used in the intervention group as follows: beginning in anesthetic induction after obtaining venous access at 1mcg/kg/h for 20 minutes, followed by 0.2 - 0.5 mcg/kg/h until surgery was completed. The placebo group will receive 0.9% saline infusion at the same rates as the intervention group. Venous blood samples were collected at three times (T1, T2 and T3): Before anesthetic induction with collection in the preoperative environment on the day of surgery or during venoclysis before anesthetic induction (sample 1, T1); 6 hours after starting orifice closure and completion of drug or placebo infusion (sample 2, T2); and the last blood sample will be collected by me on the morning after the postoperative period, close to hospital discharge (sample 3, T3). Will be measured in all venous blood samples: IL-6, cortisol, CRP and glycemia (dosing techniques -chemiluminescence or ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I and II
* Elective Videolaparoscopic Cholecystectomy Surgery
* Patients who signed the Free and Informed Consent Form

Exclusion Criteria:

* Patients ASA > II
* Conversion to open surgery
* Emergency Surgeries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Attenuation of the inflammatory response to trauma | Up to 24 hours
  Attenuation of the inflammatory response to trauma, with a reduction in the levels of Interleukin 6, C-Reactive Protein and cortisol, through a decrease of at least 5% in the values of the samples of the intervention group.

SECONDARY OUTCOMES:
Physiological functions more preserved than the control group | Up to 24 hours
  Postoperative analgesic and antiemetic effects, early return of physiological functions, verified by a reduction of at least 10% in pain scores; capnography greater than 40 mmHg; respiratory rate greater than 12 bpm and tidal volume of 6 to 8 mL/kg (absence of pathological changes in pulmonary function).

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Silva, MD, Principal Investigator — UNIRIO - FEDERAL UNIVERSITY OF THE STATE OF RIO DE JANEIRO
Locations (1):
- University Hospital Gaffree and Guinle, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva GN, Brandao VG, Fiorelli R, Perez MV, Mello CR, Negrini D, Levandrowski KU, Martinelli RB, Reis TPDAD. Outcomes of dexmedetomidine as adjuvant drug in patients undergoing videolaparoscopic cholecystectomy: A randomized and prospective clinical trial. Int J Immunopathol Pharmacol. 2023 Jan-Dec;37:3946320231196977. doi: 10.1177/03946320231196977. PMID 37604516